CLINICAL TRIAL: NCT06790823
Title: Effect of Probiotic Supplement on Improvement of Depressive Symptoms in Patients With Substance-Induced Depressive Disorder: A Randomized, Double-Blind, Placebo-Controlled Clinical Trial
Brief Title: Effect of Probiotic Supplement on Improvement of Depressive Symptoms in Patients With Substance-Induced Depressive Disorder
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Shiraz University of Medical Sciences (Other)
Responsible Party: Principal Investigator, seyed hamdollah mosavat, Clinical Professor, Shiraz University of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IR.SUMS.REC.1400.442
Record Dates: First submitted 2025-01-18; First posted 2025-01-24 (Actual); Last update posted 2025-06-13 (Actual); Status verified 2025-06

CONDITIONS: Depressive Disorder; Depressive Disorder, Major Depressive Disorder
MeSH Terms: conditions — Depressive Disorder; Depressive Disorder, Major

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Probiotic (Active Comparator): Participants were asked to take two capsules per day for four weeks, preferably before a meal.
  Interventions: Drug: The probiotic supplement (Moodamin capsuls)
- Placebo (Placebo Comparator): Participants were asked to take two placebo capsules per day for four weeks, preferably before a meal.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: The probiotic supplement (Moodamin capsuls) — The probiotic supplement (Moodamin capsuls) provided from Amin pharmacytical company, Iran, was freeze-dried containing Lactobacillus helveticus and Bifidobacterium Longum bacteria at a dose of 2.682 × CFU and 0.318 × CFU each capsule, respectively.Excipients include xylitol, maltodextrin, plum flavor, and malic acid.
  Arms: Probiotic
Drug: Placebo — The probiotic supplement (Moodamin capsuls) provided from Amin pharmacytical company, Iran, was freeze-dried containing Lactobacillus helveticus and Bifidobacterium Longum bacteria at a dose of 2.682 × CFU and 0.318 × CFU each capsule, respectively. Excipients include xylitol, maltodextrin, plum flavor, and malic acid. A placebo product used for the control group was made up of excipients only.
  Arms: Placebo

SUMMARY:
This study investigates the potential of probiotics as a therapeutic intervention for Substance-Induced Depressive Disorder (SIDD). The primary question the study aims to answer is: Can a four-week course of probiotics improve depressive symptoms and alter immune markers in patients diagnosed with SIDD, compared to a placebo?

The study uses a double-blind, placebo-controlled, randomized clinical trial design with 40 participants to explore this question by measuring clinical outcomes using BDI and HAM-A and immunological markers.

ELIGIBILITY:
Inclusion Criteria:

* Males and females, aged between 18 and 70 years
* Diagnosis of Substance-Induced Depressive Disorder as per DSM-5 criteria
* Absence of significant internal diseases as per exclusion criteria

Exclusion Criteria:

* Pregnant or lactating
* Patients who for any reason cannot comply with adequate follow-up

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2022-07-15 (Actual); Primary Completion 2023-04-12 (Actual); Study Completion 2023-04-12 (Actual)

PRIMARY OUTCOMES:
The Beck Depression Severity | 4 weeks
  The Beck Depression Severity Questionnaire used to assess the severity of depressive symptoms in participants.

CONTACTS AND LOCATIONS:
Locations (1):
- Shiraz University of Medical Sciences, Shiraz, Iran, Shiraz, Fars, Iran

IPD SHARING:
Plan to Share IPD: Undecided